CLINICAL TRIAL: NCT02871921
Title: Internet-based Conversational Engagement Clinical Trial
Acronym: I-CONECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Michigan (Other); National Institute on Aging (NIA) (NIH); Wayne State University (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Hiroko Hayama Dodge, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023p000367; R56AG056102 (NIH); R01AG051628 (NIH); R01AG056102 (NIH)
Record Dates: First submitted 2016-08-08; First posted 2016-08-18 (Estimated); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Aging; Mild Cognitive Impairment
Keywords: Behavioral intervention; social interaction; social isolation; loneliness; dementia, cognitive decline; MRI/fMRI; objective IADL assessment; speech characteristics (acoustic and linguistic); emotional well-being
MeSH Terms: conditions — Cognitive Dysfunction; Social Isolation; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study assessors will be blinded to the subject study arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversational Engagement (Experimental): Participants engage in 30-minute face-to-face communications with study staff through internet/webcam 4 times per week for 24 weeks (6 months). Under an exploratory aim, a limited number of participants will be further followed by sustaining dose of 2 times per week of 30 minutes session for additional 24 weeks (6 months). Conversational staff will facilitate content-standardized but naturalistic-style social engagement. Staff and participants will engage in conversation about a wide variety of topics that are culturally and personally relevant and interesting to participants. Each day, participants will be able to choose from topic options. Participants will also receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participant social activities and health conditions.
  Interventions: Behavioral: Conversational Engagement
- Control Group (No Intervention): Participants will receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participant social activities and health conditions

INTERVENTIONS:
Behavioral: Conversational Engagement — Examine whether increasing social interaction through face-to-face (video chat) conversations could improve cognitive function and whether the efficacy is mediated by improved psychological well-being, targeting older adults aged 75 and older who are socially isolated
  Arms: Conversational Engagement

SUMMARY:
The study aims to randomize 320 (160 Caucasian, 160 African American) socially isolated adults 75+ years old (50:50 split between those with normal cognition and mild cognitive impairment (MCI)) recruited from the community to either the Video Chat Group or the Control Group. The participants in the Video Chat Group will receive a computer and internet service for the duration of the study, which they will use to video chat with study staff for 30 minutes/day 4x/week for 6 months (high dose), and then 2x/week for an additional 6 months (maintenance dose). The efficacy examination of the maintenance dose is limited to an exploratory aim. Both intervention and control groups will have a brief (about 10 minutes) telephone check-in with study staff once per week. In-home testing will occur at Baseline and 6 months. A sub-sample of participants** will be assessed at 12 months (exploratory) after additional 6 months of maintenance dose. All participants at OHSU will have their medication compliance tracked using an electronic medication monitoring device and participants at both OHSU and UM will have MRIs at Baseline and 6 months, if they are able to safely receive MRIs. Participants at both sites will contribute saliva for genetic testing (optional consent), and all video chat and neuropsychological assessment sessions will be recorded for speech and language analysis (consent required for participation).

DETAILED DESCRIPTION:
**Due to COVID-19 pandemic and resultant research hiatus and the subsequent changes in assessment modality from in-person to telephone (T-COG) assessments, M12 (Months 12) assessments are conducted only among those who completed M12 assessments before March, 18, 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Age 75 or older
2. Consent to MRI (if physically able to receive one)
3. Socially isolated, defined by at least one of the following:

   i. Score ≤12 on the 6-item Lubben Social Network Scale (LSNS-6), ii. Engages in conversations lasting 30 minutes or longer no more than twice per week, per subject self-report iii. Answers "Often" to at least one question on the Hughes et al. Three-Item Loneliness Scale
4. Adequate vision to use study technology and complete all neuropsychological tests throughout the study, defined by the following two criteria:

   i. See well enough to complete the MoCA ii. See well enough to read a newspaper, wearing glasses if needed but not using a magnifying glass
5. Adequate hearing to use study technology and complete all neuropsychological tests throughout the study, defined as i. Able to hear well enough to complete the telephone screening ii. Able to hear well enough to complete the MoCA
6. Sufficient ability to understand English in order to complete protocol-required testing
7. Normal cognition or mild cognitive impairment (MCI), as assessed by the trial neuropsychologist
8. Sufficiently able to comply with protocol assessments and procedures, in the opinion of the investigator

Exclusion Criteria:

1. Identified as having dementia based on either of the following criteria:

   i. Self-reported diseases associated with dementia, such as Alzheimer's disease, vascular dementia, Lewy body dementia, front temporal dementia, normal pressure hydrocephalus, or Parkinson's disease ii. Diagnosis of dementia by trial neuropsychologist
2. Anticipating major change in living arrangement within the upcoming year
3. Severely depressed, operationally defined as a 15-item GDS score > 7
4. Significant disease of the central nervous system, such as brain tumor, seizure disorder, subdural hematoma, or significant stroke, per subject report
5. Current (within 2 years of screening) alcohol or substance abuse
6. Unstable or significantly symptomatic psychiatric disorder, such as major depression, schizophrenia, posttraumatic stress disorder, or bipolar disorder
7. Unstable or significantly symptomatic cardiovascular disease, such as coronary artery disease with frequent angina, or congestive heart failure with shortness of breath at rest
8. Unstable insulin-dependent diabetes mellitus, defined as meeting any of the following criteria:

   i. Received a diagnosis of Type 1 Diabetes ii. Started taking insulin within 3 months of the screening visit iii. Been hospitalized for hypoglycemia within one year of screening
9. Active systemic cancer within 5 years of the screening visit (Gleason Grade < 3 prostate cancer and non-metastatic skin cancers are acceptable)
10. Surgery that required full sedation with intubation within 6 months of screening (sedation for minor procedures is acceptable)
11. More than one overnight hospital stay within 3 months of the screening visit
12. Any other condition that, in the opinion of the investigator, is severe enough to cause study participation to have a negative impact on participant or study team rights or wellbeing.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 186 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroko Dodge, PhD, Principal Investigator — Oregon Health and Science Univeristy
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
All de-identified subject data will stored in a data repository at the conclusion of the research, and made available to approved investigators per a repository protocol.
Time Frame: Data will be available once main trial analyses have concluded, and will be available indefinitely.
Access Criteria: Investigators may access trial data via a repository data sharing request process. Data access will be granted to achieve the aims as outlined in approved data requests. IRB approval may be required.

REFERENCES:
- [Background] Yu K, Wild K, Potempa K, Hampstead BM, Lichtenberg PA, Struble LM, Pruitt P, Alfaro EL, Lindsley J, MacDonald M, Kaye JA, Silbert LC, Dodge HH. The Internet-Based Conversational Engagement Clinical Trial (I-CONECT) in Socially Isolated Adults 75+ Years Old: Randomized Controlled Trial Protocol and COVID-19 Related Study Modifications. Front Digit Health. 2021 Aug 25;3:714813. doi: 10.3389/fdgth.2021.714813. eCollection 2021. PMID 34713183
- [Background] Tang F, Chen J, Dodge HH, Zhou J. The Joint Effects of Acoustic and Linguistic Markers for Early Identification of Mild Cognitive Impairment. Front Digit Health. 2022 Feb 11;3:702772. doi: 10.3389/fdgth.2021.702772. eCollection 2021. PMID 35224534
- [Background] Liu G, Xue Z, Zhan L, Dodge HH, Zhou J. Detection of Mild Cognitive Impairment from Language Markers with Crossmodal Augmentation. Pac Symp Biocomput. 2023;28:7-18. PMID 36540960
- [Background] Chen L, Dodge HH, Asgari M. Topic-Based Measures of Conversation for Detecting Mild Cognitive Impairment. Proc Conf Assoc Comput Linguist Meet. 2020 Jul;2020:63-67. PMID 33642674
- [Background] Wu CY, Mattek N, Wild K, Miller LM, Kaye JA, Silbert LC, Dodge HH. Can changes in social contact (frequency and mode) mitigate low mood before and during the COVID-19 pandemic? The I-CONECT project. J Am Geriatr Soc. 2022 Mar;70(3):669-676. doi: 10.1111/jgs.17607. Epub 2021 Dec 13. PMID 34881436
- [Background] Yu K, Wild K, Dowling NM, Kaye JA, Silbert LC, Dodge HH. Emotional characteristics of socially isolated older adults with MCI using tablet administered NIH toolbox: I-CONECT study. Alzheimers Dement (Amst). 2022 Nov 11;14(1):e12372. doi: 10.1002/dad2.12372. eCollection 2022. PMID 36381558
- [Result] Dodge HH, Yu K, Wu CY, Pruitt PJ, Asgari M, Kaye JA, Hampstead BM, Struble L, Potempa K, Lichtenberg P, Croff R, Albin RL, Silbert LC; I-CONECT Team. Internet-Based Conversational Engagement Randomized Controlled Clinical Trial (I-CONECT) Among Socially Isolated Adults 75+ Years Old With Normal Cognition or Mild Cognitive Impairment: Topline Results. Gerontologist. 2024 Apr 1;64(4):gnad147. doi: 10.1093/geront/gnad147. PMID 37935416
- [Derived] Wu CY, Chen L, Dickson JR, Zhang B, Arnold SE, Dodge HH. Synthetic control methods for n-of-1 and parallel-group trials in Alzheimer's disease: A proof-of-concept study using the I-CONECT. Alzheimers Dement. 2025 Jul;21(7):e70460. doi: 10.1002/alz.70460. PMID 40621876
- [Derived] Yuan F, Zhou W, Dodge HH, Zhao X. Short: Causal structural learning of conversational engagement for socially isolated older adults. Smart Health (Amst). 2023 Jun;28:100384. doi: 10.1016/j.smhl.2023.100384. Epub 2023 Mar 21. PMID 37065441
- See also: Study Website — http://www.i-conect.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted between July 2018 and December 2020 from Portland, Oregon, and Detroit, Michigan; Potential subjects were identified via publicly available data; word-of-mouth referrals, and registries.
Pre-assignment Details: 2 arms were pre-assigned: Conversational Engagement vs Control Group; and were later analyzed by Cognitive Status (Normal Cognition vs MCI).
Groups:
- Conversational Engagement (MCI); Conversational Engagement (NC): Participants engage in 30-minute face-to-face communications with study staff through internet/webcam 4 times per week for 24 weeks (6 months). Under an exploratory aim, a limited number of participants will be further followed by sustaining dose of 2 times per week of 30 minutes session for additional 24 weeks (6 months). Conversational staff will facilitate content-standardized but naturalistic-style social engagement. Staff and participants will engage in conversation about a wide variety of topics that are culturally and personally relevant and interesting to participants. Each day, participants will be able to choose from topic options. Participants will also receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participant social activities and health conditions.
  Conversational Engagement: Examine whether increasing social interaction through face-to-face (video chat) conversations could improve cognitive function and whether the efficacy is mediated by improved psychological well-being, targeting older adults aged 75 and older who are socially isolated
- Control Group (MCI): Participants receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participants' social activities and health conditions
- Control Group (NC): Participants will receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participant social activities and health conditions
Period: Overall Study
Arm/Group | Conversational Engagement (MCI) | Control Group (MCI) | Control Group (NC) | Conversational Engagement (NC)
Started | 51 | 49 | 43 | 43
Month 6 | 33 | 41 | 36 | 31
Month 12 | 18 | 22 | 17 | 14
Completed | 17 | 22 | 16 | 13
Not Completed | 34 | 27 | 27 | 30
Not completed — Withdrawal by Subject | 34 | 27 | 27 | 30

BASELINE CHARACTERISTICS:
Groups:
- Control Group (MCI): Participants will receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participant social activities and health conditions
- Total: Total of all reporting groups
Arm/Group | Conversational Engagement (NC) | Control Group (NC) | Conversational Engagement (MCI) | Control Group (MCI) | Total
Number analyzed (Participants) | 43 | 43 | 51 | 49 | 186
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 79.6 (4) | 80 (3.7) | 81.9 (4.9) | 82.6 (4.9) | 81 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 34 | 31 | 130
  Male | 13 | 8 | 17 | 18 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 43 | 51 | 49 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 13 | 10 | 35
  White | 37 | 36 | 37 | 39 | 149
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intervention Efficacy for High Dose : Global Cognitive Function as Calculated From the Change From Baseline to Month 6
Description: Global cognitive function measured by the Montreal Cognitive Assessment total score (MoCA total score). Montreal Cognitive Assessment is a neuropsychological test. Total score ranges from 0 to 30. Higher scores indicate better cognitive function.
Time Frame: Change from baseline to month 6
Population: The pre-pandemic cohort consists of participants who received in-person assessments both at baseline and M6 assessments using the MoCA full battery. During the COVID-19 pandemic, telephone MoCA was used. In the pre-and post-pandemic combined cohort, missing items in telephone MoCA were imputed using available test items. The final report shows model-based analysis results that controlled for confounders.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conversational Engagement (NC) | Control Group (NC) | Conversational Engagement (MCI) | Control Group (MCI)
Number analyzed (Participants) | 31 | 35 | 33 | 41
units on a scale
  Pre-pandemic cohort MoCA | 0.40 (2.27) | 0.07 (2.34) | 1.46 (2.11) | -0.44 (2.04)
  Pre- and post-pandemic combined cohorts combined | -0.28 (2.30) | 0.31 (2.25) | 1.37 (3.04) | 0.22 (2.33)
Statistical Analysis 1: Comparison: Conversational Engagement (NC) vs Control Group (NC); Outcome: MoCA at Month 6 Among participants with normal cognition; Test type: Equivalence — A linear regression model was run with the outcome being the MoCA score at Month 6, controlling for the baseline MoCA score. The coefficient of the treatment indicator (1: experimental group, 0: control group) is our main interest. The significant coefficient means that treatment and control groups differ in the outcome score at Month 6, controlling for the baseline score; p = 0.87, Regression, Linear; Mean Difference (Final Values) = 0.14, Standard Error of Mean .86
Statistical Analysis 2: Comparison: Conversational Engagement (MCI) vs Control Group (MCI); Outcome: MoCA at Month 6 Among MCI; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .03, Regression, Linear; Mean Difference (Final Values) = 1.75, Standard Error of Mean 0.76

2. Secondary Outcome: Intervention Efficacy for High Dose: Language-based Executive Function
Description: Cognitive function in language-based executive function measured by Verbal Fluency Animal test. Verbal fluency Animals test is a neuropsychological test. In the test, participants have to produce as many words as possible from a category of animals within 60 seconds. Total score ranges from 0 to 70. Higher scores indicate better cognitive function.
Time Frame: Change from baseline to month 6
Population: Pre- and post-pandemic cohorts combined, participants with both baseline and M6 assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conversational Engagement (NC) | Control Group (NC) | Conversational Engagement (MCI) | Control Group (MCI)
Number analyzed (Participants) | 31 | 35 | 33 | 41
score on a scale | 1.06 (4.24) | -0.46 (4.30) | -0.42 (3.96) | -0.59 (4.11)
Statistical Analysis 1: Comparison: Conversational Engagement (NC) vs Control Group (NC); Outcome: Category fluency animals Among participants with normal cognition; Test type: Equivalence — A linear regression model was run with the outcome being the Category Fluency test score at Month 6, controlling for tits baseline score. The coefficient of the treatment indicator (1: experimental group, 0: control group) is our main interest. The significant coefficient means that treatment and control groups differ in the outcome score at Month 6, controlling for the baseline score and a COVID-19 pandemic period indicator (0: pre-COVID-19 pandemic, 1: during COVID-19 pandemic period); p = 0.03, Regression, Linear; Mean Difference (Final Values) = 2.56, Standard Error of Mean 1.19
Statistical Analysis 2: Comparison: Conversational Engagement (MCI) vs Control Group (MCI); Outcome: Category Fluency (Animals) at Month 6 Among MCI participants; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.46, Regression, Linear; Mean Difference (Final Values) = 0.69, Standard Error of Mean 0.93

3. Secondary Outcome: Intervention Efficacy for High Dose: Learning Function
Description: Cognitive function in a learning domain (immediate recall) measured by Craft Story Immediate Recall test (paraphrase scoring). Craft Story Immediate Recall test (paraphrase scoring) is a neuropsychological test. Total score ranges from 0 to 25. Higher scores indicate better cognitive function. Scores reported are the mean change in score.
Time Frame: Change from baseline to month 6
Population: Pre- and post-pandemic cohorts combined, participants with both baseline and M6 assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conversational Engagement (NC) | Control Group (NC) | Conversational Engagement (MCI) | Control Group (MCI)
Number analyzed (Participants) | 31 | 35 | 33 | 41
units on a scale | -.58 (3.58) | .63 (3.45) | .73 (3.51) | .95 (3.76)
Statistical Analysis 1: Comparison: Conversational Engagement (NC) vs Control Group (NC); Outcome: Craft Stroy Immediate Recall (paraphrase scoring) Among participants with normal cognition; Test type: Equivalence — A linear regression model was run with the outcome being the Craft Stroy Immediate Recall score at Month 6, controlling for its baseline score. The coefficient of the treatment indicator (1: experimental group, 0: control group) is our main interest. The significant coefficient means that treatment and control groups differ in the outcome score at Month 6, controlling for the baseline score and a COVID-19 pandemic period indicator (0: pre-COVID-19 pandemic, 1: during COVID-19 pandemic period); p = 0.45, Regression, Linear; Mean Difference (Final Values) = -0.63, Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Conversational Engagement (MCI) vs Control Group (MCI); Outcome: Craft Story Immediate Recall (paraphrase) Among MCI; Test type: Equivalence — A linear regression model was run with the outcome being the Craft Story score at Month 6, controlling for tits baseline score. The coefficient of the treatment indicator (1: experimental group, 0: control group) is our main interest. The significant coefficient means that treatment and control groups differ in the outcome score at Month 6, controlling for the baseline score and a COVID-19 pandemic period indicator (0: pre-COVID-19 pandemic, 1: during COVID-19 pandemic period); p = 0.41, Regression, Linear; Mean Difference (Final Values) = -0.66, Standard Error of Mean .80

4. Secondary Outcome: Intervention Efficacy for High Dose: Memory Function
Description: Cognitive function in a memory domain measured by Craft Story Delayed Recall test scores (paraphrase scoring). Craft Story Delayed Recall test (paraphrase scoring) is a neuropsychological test. Total score ranges from 0 to 25. Higher scores indicate better cognitive function. Scores are reported as a change score.
Time Frame: Change from baseline to month 6
Population: Pre- and post-pandemic cohorts combined, participants with both baseline and M6 assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conversational Engagement (NC) | Control Group (NC) | Conversational Engagement (MCI) | Control Group (MCI)
Number analyzed (Participants) | 31 | 35 | 33 | 40
units on a scale | -.26 (3.88) | .74 (3.37) | 1.48 (4.47) | 1.08 (3.56)
Statistical Analysis 1: Comparison: Conversational Engagement (NC) vs Control Group (NC); Outcome: Craft Story Delayed Recall) (Paraphrase scoring) Among participants with normal cognition; Test type: Equivalence — A linear regression model was run with the outcome being the Craft Story test score at Month 6, controlling for tits baseline score. The coefficient of the treatment indicator (1: experimental group, 0: control group) is our main interest. The significant coefficient means that treatment and control groups differ in the outcome score at Month 6, controlling for the baseline score and a COVID-19 pandemic period indicator (0: pre-COVID-19 pandemic, 1: during COVID-19 pandemic period); p = 0.74, Regression, Linear; Median Difference (Final Values) = -0.26, Standard Error of Mean .77
Statistical Analysis 2: Comparison: Conversational Engagement (MCI) vs Control Group (MCI); Outcome: Craft Story Delayed Recall (Paraphrase scoring) Among MCI; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.90, Regression, Linear; Median Difference (Final Values) = -0.10, Standard Error of Mean .79

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 2 years, from baseline to follow-up.
Description: 2 Arms were analyzed for Adverse Events (Conversational Engagement vs Control Group).
Groups:
- Control Group(NC): Participants will receive a phone call once per week that lasts approximately 10 minutes; interviewers ask brief questions to monitor participant social activities and health conditions
Arm/Group | Conversational Engagement (MCI) | Control Group (MCI) | Conversational Engagement (NC) | Control Group(NC)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 2/51 | 0/49 | 0/43 | 1/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conversational Engagement (MCI) (N=51) | Control Group (MCI) (N=49) | Conversational Engagement (NC) (N=43) | Control Group(NC) (N=43)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02871921/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02871921/ICF_001.pdf